CLINICAL TRIAL: NCT06746402
Title: A Phase 1, Two-Part, Double-blind, Placebo-controlled, Randomized Study of the Safety, Tolerability, and Pharmacokinetics of BMS-986278 (Part A) and a Randomized, Double-blind, Positive-controlled, Placebo-controlled, 4-Period Crossover, Thorough QT/QTc Study to Evaluate the Effect of Multiple Doses of BMS-986278 on Cardiac Repolarization (Part B) in Healthy Participants
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of BMS-986278 and the Effects of BMS-986278 on Cardiac Repolarization in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM027-1012
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Part A, a parallel model, will be followed by Part B, a 4-way crossover model.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study, with an open-label positive control in Part B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A (Experimental)
  Interventions: Drug: BMS-986278; Drug: Placebo
- Part B1/B2 Treatment A (Experimental)
  Interventions: Drug: BMS-986278
- Part B1/B2 Treatment B (Experimental)
  Interventions: Drug: BMS-986278; Drug: Placebo
- Part B1/B2 Treatment C (Experimental)
  Interventions: Drug: Placebo
- Part B1/B2 Treatment D (Experimental)
  Interventions: Drug: Placebo; Drug: Moxifloxacin
- Part B3 Treatment A (Experimental)
  Interventions: Drug: BMS-986278
- Part B3 Treatment B (Experimental)
  Interventions: Drug: BMS-986278; Drug: Placebo
- Part B3 Treatment C (Experimental)
  Interventions: Drug: Placebo
- Part B3 Treatment D (Experimental)
  Interventions: Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days
  Arms: Part A; Part B1/B2 Treatment A; Part B1/B2 Treatment B; Part B3 Treatment A; Part B3 Treatment B
Drug: Placebo — Specified dose on specified days
  Arms: Part A; Part B1/B2 Treatment B; Part B1/B2 Treatment C; Part B1/B2 Treatment D; Part B3 Treatment B; Part B3 Treatment C; Part B3 Treatment D
Drug: Moxifloxacin — Specified dose on specified days
  Arms: Part B1/B2 Treatment D; Part B3 Treatment D

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics (PK) of high dose of BMS-986278 in healthy participants and to assess the effect of BMS-986278 on the ECG intervals in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals not of childbearing potential (INOCBP) and males.
* Healthy as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory assessments.
* Body mass index (BMI) 18.0 to 32.0 kg/m2 , inclusive, for Parts A and B.

Exclusion Criteria:

* Any significant acute or chronic medical illness as determined by the investigator.
* History of clinically relevant cardiac disease as determined by the investigator, symptomatic or asymptomatic arrhythmias, presyncope or syncopal episodes, or additional risk factors for ventricular arrhythmias.
* Any significant history of disease of the cardiovascular system that in the opinion of the Investigator makes the participant unsuitable for enrollment into the study.
* Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with non-serious Adverse Events (AEs) | Until 28 days post last treatment dose
  Part A
Number of participants with Serious AEs (SAEs) | Until 28 days post last treatment dose
  Part A
Number of participants with AEs leading to study intervention discontinuation | Until 28 days post last treatment dose
  Part A
Number of participants with vital sign abnormalities | Up to Day 18
  Part A
Number of participants with clinical laboratory assessment abnormalities | Up to Day 18
  Part A
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to Day 18
  Part A
Number of participants with physical examination abnormalities | Up to Day 18
  Part A
Change from baseline Fridericia's corrected QT interval (QTcF) (ΔQTcF) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Placebo-corrected change from baseline QTcF (ΔΔQTcF) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part A and Part B
Time of maximum observed plasma concentration (Tmax) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part A and Part B
Area under the plasma concentration-time curve from time zero to the end of dosing interval AUC(TAU) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part A and Part B
Terminal half-life (T-HALF) | Up to Day 18
  Part A
Apparent total body clearance (CLT/F) | Up to Day 18
  Part A
Change from baseline heart rate (HR) (∆HR) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Change from baseline PR interval (∆PR) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Change from baseline QRS interval (∆QRS) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Placebo-corrected change from baseline HR (ΔΔHR) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Placebo-corrected Change from baseline PR interval (ΔΔPR) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Placebo-corrected change from baseline QRS interval (ΔΔQRS) | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Number of participants with categorical outliers for QTcF | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Number of participants with categorical outliers for HR | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Number of participants with categorical outliers for PR interval | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Number of participants with categorical outliers for QRS interval | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Number of participants with treatment-emergent changes of ECG morphology | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
ΔQTcF for moxifloxacin | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
ΔΔQTcF for moxifloxacin | Up to Day 13 of Period 4 (Each period is 17 days)
  Part B
Number of participants with non-serious AEs | Until 28 days post last treatment dose
  Part B
Number of participants with SAEs | Until 28 days post last treatment dose
  Part B
Number of participants with AEs leading to study intervention discontinuation | Until 28 days post last treatment dose
  Part B
Number of participants with vital sign abnormalities | Up to Day 18 of Period 4 (Each period is 17 days)
  Part B
Number of participants with clinical laboratory assessment abnormalities | Up to Day 17 of Period 4 (Each period is 17 days)
  Part B
Number of participants with 12-lead ECG abnormalitie | Up to Day 17 of Period 4 (Each period is 17 days)
  Part B
Number of participants with physical examination abnormalities | Up to Day 18 of Period 4 (Each period is 17 days)
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - ICON San Antonio, San Antonio, Texas
  - Local Institution - 0001, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com